CLINICAL TRIAL: NCT00100789
Title: A Phase II Study of Biweekly Gemcitabine and Paclitaxel (GEMTAX) Combination in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: S0329, Gemcitabine and Paclitaxel in Treating Patients With Persistent, Recurrent, or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000407644; S0329 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-08

CONDITIONS: Head and Neck Cancer
Keywords: Recurrent; stage IV; squamous cell carcinoma; hypopharynx; larynx; lip; oral cavity; nasopharynx; oropharynx; paranasal; nasal cavity; metastatic; neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence; Carcinoma, Squamous Cell; Laryngeal Diseases; Lymphoid Interstitial Pneumonia; Neoplasm Metastasis | interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine paclitaxel combination (Experimental)
  Interventions: Drug: gemcitabine; Drug: paclitaxel

INTERVENTIONS:
Drug: gemcitabine — 3,000 mg/m2 IV over 30 minutes on days 1 and 15 (q28 days).
  Other Names: Gemzar; NSC-613327
Drug: paclitaxel — 150 mg/m2 IV over 1 hour on days 1 and 15 (q 28 day cycle), administered after gemcitabine
  Other Names: Taxol; NSC-673089

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gemcitabine together with paclitaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with paclitaxel works in treating patients with persistent, recurrent, or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine overall and progression-free survival probability in patients with persistent, recurrent, or metastatic squamous cell carcinoma of the head and neck treated with gemcitabine and paclitaxel.
* Determine the confirmed and unconfirmed response (partial and complete) probability in patients with measurable disease treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes and paclitaxel IV over 1 hour on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 4 additional courses beyond CR.

Patients are followed every 8 weeks until disease progression, every 6 month for 2 years, and then annually for 1 year.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study within 10-13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck (SCCHN)

  * Recurrent, persistent, or newly diagnosed metastatic disease
* Measurable or non-measurable disease
* No active or prior CNS metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No serious organ dysfunction
* No serious comorbid conditions that would preclude study treatment
* No history of hypersensitivity reaction to products containing polysorbate 80
* No active infection requiring systemic antibiotic therapy
* No symptomatic sensory neuropathy ≥ grade 2
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic or immunotherapy for SCCHN
* No concurrent gene therapy for SCCHN

Chemotherapy

* No prior chemotherapy for recurrent or newly diagnosed metastatic disease
* At least 6 months since prior induction or adjuvant chemotherapy

  * No more than 1 prior induction or adjuvant regimen
* No prior gemcitabine or taxanes as part of induction, adjuvant, or neoadjuvant chemotherapy
* No other concurrent chemotherapy for SCCHN

Endocrine therapy

* Not specified

Radiotherapy

* At least 28 days since prior radiotherapy and recovered
* No concurrent radiotherapy for SCCHN

Surgery

* Not specified

Other

* No other concurrent therapy for SCCHN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (123):
- United States (123):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Center for Cancer Medicine and Blood Disorders, PA, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Paclitaxel: Patients received Gemcitabine 3,000 mg/m2 (IV on days 1 and 15 over 30 minutes) and Paclitaxel 150 mg/m2 (IV on days 1 and 15 over one hour). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 4 additional courses beyond CR.
Period: Overall Study
Arm/Group | Gemcitabine and Paclitaxel
Started | 67
Eligible | 64
Eligible and Began Protocol Therapy | 63
Completed | 3
Not Completed | 64
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 1
Not completed — Progression/relapse | 42
Not completed — Death | 2
Not completed — Not protocol specified | 5
Not completed — Ineligible | 3
Not completed — Never received treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine and Paclitaxel: Patients received Gemcitabine 3,000 mg/m2 (IV on days 1 and 15 over 30 minutes) and Paclitaxel 150 mg/m2 (IV on days 1 and 15 over one hour). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 4 additional courses beyond CR. Eligible patients who received any treatment were included in baseline measures.
Arm/Group | Gemcitabine and Paclitaxel
Number analyzed (Participants) | 63
Age Continuous [Median (Full Range); unit: years] | 63.1 [40.7 to 82.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 50
  More than one race | 1
  Unknown or Not Reported | 1
Primary Site [Number; unit: participants]
  Lip/Oral Cavity | 20
  Nasopharynx | 4
  Oropharynx | 13
  Salivary glands | 0
  Hypopharynx | 2
  Larynx | 16
  Paranasal Sinuses | 3
  Other/Unknown | 5
Disease Status [Number; unit: participants]
  Newly Diagnosed | 5
  Persistent | 7
  Recurrent | 50
  Not Reported | 1
Performance Status [Number; unit: participants] — Performance status is graded according to the Zubrod Performance Status Scale. Patients with a performance status of 0 are fully active, able to carry on all pre-disease performance without restriction. Patients with a performance status of 1 are restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  participants
    0 | 24
    1 | 39

OUTCOME MEASURES:

1. Secondary Outcome: Progression-free Survival
Description: Measured from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: 0 - 3 years
Population: All eligible patients who started treatment were included in this measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Paclitaxel
Number analyzed (Participants) | 63
months | 4 [3 to 6]

2. Primary Outcome: Overall Survival
Description: Measured from time of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: 0 - 3 years
Population: All eligible patients who started treatment were included in this measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Paclitaxel
Number analyzed (Participants) | 63
months | 8 [7 to 12]

3. Secondary Outcome: Response
Description: Complete Response (CR) is complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Normalization of markers and other normal lab values. Partial Response (PR) is greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Confirmation of CR or PR means a repeat scan at least 4 weeks apart documented before progression or symptomatic deterioration.
Time Frame: 9 weeks - 3 years
Population: All eligible patients with measurable disease who started treatment were included in response measures.
Measure: Number; unit: participants
Arm/Group | Gemcitabine and Paclitaxel
Number analyzed (Participants) | 57
participants
  Complete Response | 1
  Partial Response | 6
  Unconfirmed Complete Response | 1
  Unconfirmed Partial Response | 8
  Stable/No Response | 11
  Increasing Disease | 21
  Assessment Inadequate | 9

4. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events after the first cycle of treatment and then every three months while on treatment.
Population: Eligible patients who received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants with a given type of AE
Arm/Group | Gemcitabine and Paclitaxel
Number analyzed (Participants) | 63
Participants with a given type of AE
  Allergic reaction/hypersensitivity | 1
  Anorexia | 1
  Dehydration | 1
  Diarrhea | 2
  Dyspnea (shortness of breath) | 2
  Fatigue (asthenia, lethargy, malaise) | 8
  Febrile neutropenia | 3
  Glucose, serum-high (hyperglycemia) | 1
  Hemoglobin | 2
  Hemorrhage, pulmonary/upper respiratory - Nose | 1
  Hypotension | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Catheter | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1
  Leukocytes (total WBC) | 2
  Lymphopenia | 3
  Memory impairment | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 1
  Muscle weakness, not d/t neuropathy - body/general | 1
  Neuropathy: motor | 1
  Neuropathy: sensory | 3
  Neutrophils/granulocytes (ANC/AGC) | 7
  Pain - Bone | 1
  Pain-Other (Specify) | 1
  Platelets | 2
  Pneumonitis/pulmonary infiltrates | 1
  Rash/desquamation | 1
  Rash: acne/acneiform | 1
  Sodium, serum-low (hyponatremia) | 3
  Thrombosis/thrombus/embolism | 1
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after the first cycle of treatment and then every three months while on treatment.
Arm/Group | Gemcitabine and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 54/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Paclitaxel (N=63)
Hemoglobin (Blood and lymphatic system disorders) | 41
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 6
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 10
Edema: limb (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 40
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 11
Rigors/chills (General disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 21
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 16
Alkaline phosphatase (Investigations) | 11
Leukocytes (total WBC) (Investigations) | 19
Lymphopenia (Investigations) | 19
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 17
Platelets (Investigations) | 8
Weight loss (Investigations) | 9
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 12
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 16
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7
Dizziness (Nervous system disorders) | 6
Neuropathy: motor (Nervous system disorders) | 4
Neuropathy: sensory (Nervous system disorders) | 20
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 24
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No